CLINICAL TRIAL: NCT00724828
Title: An Evaluation of Streptococcus Pneumoniae Serotype Carriage Rate For Nasopharyngeal Carriage in Filipino Children Attending Well Baby Clinic in Hospitals and Primary Care Centers
Brief Title: Study Evaluating Streptococcus Pneumoniae Serotype Carriage Rate for Nasopharyngeal Carriage in Filipino Children
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 0887X-101959
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Pneumonia, Bacterial
Keywords: Bacterial otitis media; pneumoniae; sepsis; bacteremia; meningitis; Streptococcus pneumoniae carriage rate
MeSH Terms: conditions — Pneumonia, Bacterial; Sepsis; Bacteremia; Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1

SUMMARY:
Evaluation of the carriage rate of Streptococcus pneumoniae in the nasopharynx of healthy children and the carriage rate and distribution of Streptococcus pneumoniae serotypes

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged between 2 months and 5 years attending the well baby clinic in hospital.
* Informed consent obtained from parents or legal guardian.

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2005-05; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Streptococcus pneumoniae serotype carriage rate based on a nasopharyngeal swab. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer